CLINICAL TRIAL: NCT03000413
Title: Ketamine Efficacy for Acute Severe Bronchospasm in Mechanically Ventilated-critically Ill Patients: a Randomized Controlled Trial
Brief Title: Ketamine Efficacy for Acute Severe Bronchospasm in ICU: MACANUDO Trial
Acronym: MACANUDO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Wagner Luis Nedel, MD, MSc., Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42324015.0.0000.5530
Record Dates: First submitted 2016-11-18; First posted 2016-12-22 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Critical Illness; Asthma; Bronchospasm
MeSH Terms: conditions — Critical Illness; Asthma; Bronchial Spasm | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Intravenous ketamine infusion: bolus 2mg per kg and continuous infusion (2mg/kg/h)
  Interventions: Drug: Ketamine
- Fentanyl (Active Comparator): Fentanyl: bolus infusion 1μg per kg and continuous infusion (1μg/kg/h)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine — Active treatment
  Arms: Ketamine
Drug: Fentanyl
  Arms: Fentanyl

SUMMARY:
Despite few scientific evidence that could support the use of ketamine in adult patients undergoing acute bronchospasm requiring mechanical ventilation (MV), ketamine is largely employed in this setting. The aim of this study is therefore assess more definitively the real benefit of using ketamine in patients with severe bronchospasm, requiring ICU stay and need for MV in order to establish or refute the use of this drug as "standard therapy" in these cases.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute exacerbation of COPD or status asthmaticus, undergoing controlled mechanical ventilation
* acute bronchospasm, defined as airway resistance value (Rsr max) greater than 12, use of inhaled therapy with bronchodilators and systemic corticosteroids
* patients requiring the use of continuous intravenous sedation for optimization of ventilation

Exclusion Criteria:

* contraindication or history of previous adverse events with the use of the studied drugs
* other diagnostic potential Rsr increase of not causing bronchospasm (bronchial obstruction, acute respiratory distress syndrome adult, pulmonary fibrosis)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
bronchospasm improvement | 3 hours post beginning of drug infusion
  Maximal airway resistance reduction in hour 3-post beginning of drug infusion

SECONDARY OUTCOMES:
bronchospasm improvement | 24 hours post beginning of drug infusion
  Maximal airway resistance reduction in 24th hour post beginning of drug infusion
Time to weaning | Time (in days) to first spontaneous breathing trial post randomization up to 28 days
  Time (in days) to first spontaneous breathing trial post randomization up to 28 days

OTHER OUTCOMES:
Dynamic complacence improvement | 3 hours and 24 hours post beginning of drug infusion
Air trapping improvement | 3 hours and 24 hours post beginning of drug infusion
  intrinsic PEEP reduction in 3 and 24h post beginning of drug infusion
Heart rate | 3 hours and 24 hours post beginning of drug infusion
  Heart rate in 3 hours and 24h post beginning of drug infusion
Blood pressure | 3 hours and 24 hours post beginning of drug infusion
  Blood pressure variation in 3 hours and 24hours post beginning of drug infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nossa Senhora da Conceição, Porto Alegre, Brazil

REFERENCES:
- [Background] Barbas CS, Isola AM, Farias AM, Cavalcanti AB, Gama AM, Duarte AC, Vianna A, Serpa Neto A, Bravim Bde A, Pinheiro Bdo V, Mazza BF, Carvalho CR, Toufen Junior C, David CM, Taniguchi C, Mazza DD, Dragosavac D, Toledo DO, Costa EL, Caser EB, Silva E, Amorim FF, Saddy F, Galas FR, Silva GS, Matos GF, Emmerich JC, Valiatti JL, Teles JM, Victorino JA, Ferreira JC, Prodomo LP, Hajjar LA, Martins LC, Malbouisson LM, Vargas MA, Reis MA, Amato MB, Holanda MA, Park M, Jacomelli M, Tavares M, Damasceno MC, Assuncao MS, Damasceno MP, Youssef NC, Teixeira PJ, Caruso P, Duarte PA, Messeder O, Eid RC, Rodrigues RG, Jesus RF, Kairalla RA, Justino S, Nemer SN, Romero SB, Amado VM. Brazilian recommendations of mechanical ventilation 2013. Part I. Rev Bras Ter Intensiva. 2014 Apr-Jun;26(2):89-121. doi: 10.5935/0103-507x.20140017. PMID 25028944
- [Background] Rowe BH, Sevcik W, Villa-Roel C. Management of severe acute asthma in the emergency department. Curr Opin Crit Care. 2011 Aug;17(4):335-41. doi: 10.1097/MCC.0b013e328348bf09. PMID 21716106
- [Background] Heshmati F, Zeinali MB, Noroozinia H, Abbacivash R, Mahoori A. Use of ketamine in severe status asthmaticus in intensive care unit. Iran J Allergy Asthma Immunol. 2003 Dec;2(4):175-80. PMID 17301376
- [Background] Howton JC, Rose J, Duffy S, Zoltanski T, Levitt MA. Randomized, double-blind, placebo-controlled trial of intravenous ketamine in acute asthma. Ann Emerg Med. 1996 Feb;27(2):170-5. doi: 10.1016/s0196-0644(96)70319-0. PMID 8629747
- [Background] Goyal S, Agrawal A. Ketamine in status asthmaticus: A review. Indian J Crit Care Med. 2013 May;17(3):154-61. doi: 10.4103/0972-5229.117048. PMID 24082612
- [Background] Miller AC, Jamin CT, Elamin EM. Continuous intravenous infusion of ketamine for maintenance sedation. Minerva Anestesiol. 2011 Aug;77(8):812-20. PMID 21730929
- [Background] Abu-Hijleh M, El-Sameed Y, Eldridge K, Vadia E, Chiu H, Dreyfuss Z, Al Rabadi LS. Linear probe endobronchial ultrasound bronchoscopy with guided transbronchial needle aspiration (EBUS-TBNA) in the evaluation of mediastinal and hilar pathology: introducing the procedure to a teaching institution. Lung. 2013 Feb;191(1):109-15. doi: 10.1007/s00408-012-9439-z. Epub 2012 Dec 4. PMID 23208583
- [Background] Allen JY, Macias CG. The efficacy of ketamine in pediatric emergency department patients who present with acute severe asthma. Ann Emerg Med. 2005 Jul;46(1):43-50. doi: 10.1016/j.annemergmed.2005.02.024. PMID 15988425